CLINICAL TRIAL: NCT05260736
Title: Comparison of Costoclavicular Lateral, Costoclavicular Medial and Lateral Sagittal Approaches to Infraclavicular Brachial Plexus Block in Upper Extremity Surgery
Brief Title: Comparison of Costoclavicular and Paracoracoid Approaches to Infraclavicular Brachial Plexus Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/151
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Prospective, Interventional
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Costoclavicular Lateral (CL) (Active Comparator): Patients anesthetized with costoclavicular lateral infraclavicular brachial plexus block.
  Interventions: Procedure: Infraclavicular brachial plexus block
- Group Costoclavicular Medial (CM) (Active Comparator): Patients anesthetized with costoclavicular medial infraclavicular brachial plexus block.
  Interventions: Procedure: Infraclavicular brachial plexus block
- Group Lateral Sagittal (LS) (Active Comparator): Patients anesthetized with lateral sagittal infraclavicular brachial plexus block.
  Interventions: Procedure: Infraclavicular brachial plexus block

INTERVENTIONS:
Procedure: Infraclavicular brachial plexus block — Named after the anatomical site; patients will be applied infraclavicular brachial plexus block with costoclavicular lateral, costoclavicular medial or lateral sagittal approach.

SUMMARY:
Infraclavicular block has taken its place in the literature as a proven technique in the anesthetic management of upper extremity surgeries. Compared to general anesthesia; The prominent advantages of regional anesthesia are that it provides longer perioperative pain control, reduces the incidence of postoperative nausea and vomiting, reduces opioid consumption and reduces the cost of hospitalization. The widespread use of ultrasonography (USG) in the last two decades has facilitated the application of the method and allowed the investigation of different injection methods.

Regional blocks are planned according to the surgery to be performed. For anesthesia of arm, forearm and hand operations; brachial plexus can be blocked in the axillary, infraclavicular, supraclavicular or interscalene region. The infraclavicular technique, on the other hand, is roughly divided into three types: costoclavicular lateral, costoclavicular medial and paracoracoid (Lateral sagittal). The image obtained by placing the ultrasonography probe in the relevant anatomical region serves as a guide for the orientation of the peripheral block needle and performing the intervention by observing the vascular structures in the existing region provides a great advantage in terms of patient safety.

In this study, we aimed to examine 3 different infraclavicular block methods; lateral costoclavicular, medial costoclavicular and lateral sagittal (Paracoracoid) approach, in terms of ease of application and motor/sensory block efficiency. Our hypothesis is that the sensory block will begin in a shorter time with costoclavicular methods compared to the lateral sagittal method. We are also planning to compare performance difficulties (needle maneuver numbers, subjective block exertion, block performance time etc.) for each type of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective upper extremity surgeries (Arm, upper-arm and hand)

Exclusion Criteria:

* Patients with bleeding diathesis Presence of infection on the intervention site Patients requiring continous anticoagulation therapy due to the existing comorbidities Patients with history of local anesthetic allergy Pregnant patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Sensory block onset time | Up to 45 minutes.
  Separately evaluated sensorial examination for four nerves (n. medianus, n. radialis, n. ulnaris, n. musculocutaneus), a total number of 6 points is accepted as "settled sensory block". 0= absent sensory block (feels pain), 1= partial sensory block (feels touch), 2= complete sensory block (no sense). Patients will be evaluated every 5 minutes after intervention.

SECONDARY OUTCOMES:
Ideal USG guided brachial plexus cords visualization / needle pathway planning time | Up to 15 minutes
  Practitioner's ideal image acquisition time
Needle tip and shaft imaging visualization difficulty | Up to 15 minutes
  Likert Scale: 1-5 (1:very hard; 5: very easy)
Requirement of additional maneuver due to insufficient local anesthetic distribution | Up to 15 minutes
  Extra needle redirection to cover neural structure
Total procedure difficulty according to anesthesiologist | Up to 15 minutes
  Likert Scale: 1-5 (1:Very hard; 5: Very easy)
Patient number requiring rescue analgesics | Intraoperative 2-4 hours
  If a ≥ 20% increase above preinduction values in MAP or HR was observed during the perioperative period, additional fentanyl dose (1 μg/kg) was applied intravenously
Motor blockade onset time | Up to 45 minutes
  Separately evaluated motor examination for four nerves (n. medianus, n. radialis, n. ulnaris, n. musculocutaneus), a total number of 6 points is accepted as "settled motor block". 0= absent motor block (Full movement), 1= partial motor block (free movement only), 2= complete motor block (no movement). Patients will be evaluated every 5 minutes after intervention.
Time to postoperative first pain | Up to 24 hours
  Time to first intravenous analgesic administration which is requested by the patient
Patient number requiring postoperative additional analgesic | Up to 24 hours
  Number of patients who require paracetamol (15 mg/kg) and tramadol (1mg/kg) IV
Complications / Side effects | Up to 24 hours
  Possible complications related to infraclavicular block (such as vascular puncture, hematoma, pneumothorax, diaphragma palsy...)
Patient satisfaction | Up to 24 hours
  Satisfaction score: 0: very unsatisfied 3: very satisfied
Surgeon satisfaction | Up to 24 hours
  Satisfaction score: 0: very unsatisfied, 3: very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Meltem Savran Karadeniz, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bingul ES, Canbaz M, Guzel M, Salviz EA, Akalin BE, Berkoz O, Emre Demirel E, Sungur Z, Savran Karadeniz M. Comparing the clinical features of lateral and medial approaches of costoclavicular technique versus traditional lateral sagittal technique as infraclavicular brachial plexus block methods: a randomized controlled trial. BMC Anesthesiol. 2024 Jul 25;24(1):254. doi: 10.1186/s12871-024-02645-z. PMID 39054425